CLINICAL TRIAL: NCT03837418
Title: DESIGNING A PROGRAMMING LANGUAGE FOR PATIENT-ORIENTED PRESCRIPTIONS (POP-PL)
Status: Withdrawn | Type: Observational
Why Stopped: Investigator is no longer at Northwestern University.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephanie Rangel, Research Assistant Professor of Dermatology, Northwestern University
Other Study IDs: SMB03092018
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Programming Languages; Patients
Keywords: Patient-Oriented; Designing; Prescriptions
MeSH Terms: conditions — Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to create a human-readable and executable computer language to implement medical prescriptions and to evaluate and refine this language, with the goal of improving safety and efficacy of patient care

DETAILED DESCRIPTION:
Preventable errors in healthcare are a leading cause of patient injury and death. Despite extensive effort and the expenditure of billions of dollars, computerization has failed to solve this problem. Research has shown that software design and debugging of a paper prescription markedly decreases the rate of injury and death associated with use of opioids in hospitalized patients. To further the application of insights from software engineering to the practice of medicine, the PIs will design and build a Patient-Oriented Prescription Programming Language (POP-PL) and evaluate if this new platform can be used to improve medical management of patients. The design of POP-PL will be based on building an understanding of the process of medical treatment of patients. This project is a collaboration between computer scientists and clinicians at Northwestern Medicine. The collaborating clinicians are co-investigators on this research project and also are providing healthcare to the patients that are being observed. The computer scientists and other research staff have undergone human subjects research training and are co-investigators on this research project as well. The clinician-investigators will oversee research project staff during all observations of patients, clinical encounters between healthcare providers and patients, and interactions between healthcare providers and healthcare information systems. Researchers involved in this study will observe interactions between health care providers and patients and will collate these observations with data from electronic data sources. Since this research is based mainly upon observation and chart review and will not involve any interventions or changes to patient care, the risk to study participants is minimal, involving inadvertent disclosure of healthcare information. This risk will be mitigated by anonymizing collected data.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at Northwestern Memorial Hospital, Northwestern Medicine Clinics, Lurie Children's Clinics, and Lurie Children's Hospital between the ages of 0-79.

Exclusion Criteria:

* Patients without data within the NMEDW medical record database or LCH CDW or BIS medical record database.

Ages: 0 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen at Northwestern Memorial Hospital, Northwestern Medicine Clinics, Lurie Children's Clinics, and Lurie Children's Hospital between the ages of 0-79.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Differences between Ideal and Actual Performance of Prescriptions by Number of Deviations between Sequences of Events | 2 years
  Investigators will express the intent of prescriptions in prescription programming language. Investigators will then compare the actual performance of the prescription in a clinical environment to the performance of the prescription in a simulated environment based on the same inputs as occurred in the real clinical environment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Belknap, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No